CLINICAL TRIAL: NCT04626050
Title: A Brief Phased Two-Step Intervention for Treating General Psychological Distress, PTSD and Co-Morbidities in Healthcare Workers Consequent to the COVID-19 Pandemic
Brief Title: General Psychological Distress, PTSD, and Co-Morbidities in Healthcare Workers Consequent to COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 20-04021913
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Post-traumatic Stress Disorder; Moral Injury
Keywords: PTSD; Moral Injury; Psychological Distress; Healthcare Workers; COVID-19; COVID-19 Pandemic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19 | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be aware of the condition for Phase 1 or Phase 2 of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Medical Music (Phase I) (Experimental): Participants will complete four medical music sessions that are 20 minutes in length each.
  Interventions: Behavioral: Medical Music
- Narrative Writing (Phase I) (Experimental): Participants will complete four narrative writing sessions that are 20 minutes in length each.
  Interventions: Behavioral: Narrative Writing
- Interpersonal Psychotherapy (Phase II) (Active Comparator): IPT is comprised of ten 75-minute sessions scheduled twice weekly.
  Interventions: Behavioral: Interpersonal Psychotherapy
- Prolonged Exposure Therapy (Phase II) (Active Comparator): ET is comprised of ten 75-minute sessions scheduled twice weekly.
  Interventions: Behavioral: Prolonged Exposure Therapy

INTERVENTIONS:
Behavioral: Medical Music — Participants randomized to this condition will complete 4 medical music sessions over the course of 2 weeks
  Arms: Medical Music (Phase I)
Behavioral: Narrative Writing — Participants randomized to this condition will complete 4 narrative writing sessions over the course of 2 weeks
  Arms: Narrative Writing (Phase I)
Behavioral: Prolonged Exposure Therapy — Psychotherapy including imaginal exposure for PTSD
  Arms: Prolonged Exposure Therapy (Phase II)
Behavioral: Interpersonal Psychotherapy — Psychotherapy that focuses on the effects of PTSD on current interpersonal functioning
  Arms: Interpersonal Psychotherapy (Phase II)

SUMMARY:
It is expected that large numbers of healthcare workers will experience a broad range of psychological reactions and symptoms including anxiety, depression, moral distress, and trauma symptoms that will cause both significant suffering as well as occupational and social impairment. The purpose of this study is to find interventions which are helpful in treating psychological distress in healthcare workers caring for COVID-19 patients.

There are two phases of the study. All participants will take part in Phase I, which consists of 4 sessions over a two-week period of either a narrative writing intervention or a medical music intervention. Participants will be randomly assigned to the narrative writing intervention or medical music intervention.

After Phase I, participants will be re-assessed. Healthcare workers who meet criteria for PTSD will be given the option to participate in Phase II of the study, in which they will be offered a choice between one of two evidence-based treatments for PTSD: Interpersonal Therapy (IPT) or Exposure Therapy (ET). Both treatments are comprised of ten 75-minute sessions scheduled twice weekly. Participants will be allowed to choose a preferred treatment in Phase II. After Phase II participants will complete a final assessment concluding the study. All interventions will be offered using distance technology.

ELIGIBILITY:
Inclusion Criteria:

* Any healthcare worker providing medical care or support for COVID-19 patients
* English-speaking
* Age >18
* Medically stable
* Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments
* If on psychotropic medication stable for prior 60 days

For phase II additional inclusion criteria:

- Current diagnosis of PTSD

Exclusion Criteria:

* Current significant unstable medical illness precluding regular session attendance or assessment completion
* Participants who in the investigator's judgment pose a current homicidal, suicidal, or other risk
* Lifetime or current diagnosis of schizophrenia or other psychotic disorder
* Participation in a clinical trial or concurrent evidence-based treatment for psychiatric conditions or PTSD during the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator: Recruitment (Phase I) | Baseline
  Feasibility assessment will include recruitment defined as number of individuals interested in the intervention.
Feasibility Indicator: Recruitment (Phase II) | Post-Phase I Assessment at week 2
  Feasibility assessment will include: recruitment defined as number of individuals interested in the intervention.
Feasibility Indicator: Enrollment (Phase I) | Baseline
  Feasibility assessment will include enrollment defined as number of participants signing the informed consent form.
Feasibility Indicator: Enrollment (Phase II) | Post-Phase I Assessment at approximately week 2
  Feasibility assessment will include enrollment defined as number of individuals beginning phase II.
Feasibility Indicator: Retention (Phase I) | Post-Phase I Assessment at approximately week 2
  Feasibility assessment will include retention defined as the number of participants completing the full course of Phase I interventions.
Feasibility Indicator: Retention (Phase II) | Post-Phase II Assessment at approximately week 7
  Feasibility assessment will include retention defined as the number of participants completing the full course of Phase II interventions.
Acceptability Indicator: Satisfaction (Phase I) | Post-Phase I Assessment at approximately week 2
  Acceptability and treatment satisfaction will be rated with a Likert scale.
Acceptability Indicator: Satisfaction (Phase II) | Post-Phase II Assessment at approximately week 7
  Acceptability and treatment satisfaction will be rated with a Likert scale.
Preliminary Efficacy as Measured by Change in Clinician-Administered PTSD Scale Score (Phase I) | Start of Phase I to approximately 2 weeks
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score. Total Scores range from 0-80. Higher scores indicate greater symptom severity.
Preliminary Efficacy as Measured by Change in Clinician-Administered PTSD Scale Score (Phase II) | Start of Phase II to approximately 5 weeks
  Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Score. Total Scores range from 0-80. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms measured by the Generalized Anxiety Disorder 7-Item Scale (Phase I) | Start of Phase I to approximately 2 weeks
  Scored between 0-21:
  Cut offs:
  0-4 = None 5-9 = Mild anxiety 10-14 = Moderate anxiety 15-21 = Severe anxiety
  Higher scores indicate greater symptom severity.
Change in Anxiety Symptoms measured by the Generalized Anxiety Disorder 7-Item Scale (Phase II) | Start of Phase II to approximately 5 weeks
  Scored between 0-21:
  Cut offs:
  0-4 = None 5-9 = Mild anxiety 10-14 = Moderate anxiety 15-21 = Severe anxiety
  Higher scores indicate greater symptom severity.
Change in Depressive Symptoms measured by the Quick Inventory of Depressive Symptomology (Phase I) | Start of Phase I to approximately 2 weeks
  16-item self-report measure. Scored between 0-3. Higher scores indicate greater symptom severity
Change in Depressive Symptoms measured by the Quick Inventory of Depressive Symptomology (Phase II) | Start of Phase II to approximately 5 weeks
  16-item self-report measure. Scored between 0-3. Higher scores indicate greater symptom severity.
Change in score on the Pittsburgh Sleep Quality Index (PSQI) (Phase I) | Start of Phase I to approximately 2 weeks
  24 item self-report measure. 19 questions are evaluated. Each item in the scale is rated between 0 (no distress) and 3 (serious distress). The total PSQI score ranges from 0-21. Sleep quality of the patients with a total score of 5 and below is considered "good". A score of greater than 5 refers to poor sleep quality.
Change in score on the Pittsburgh Sleep Quality Index (PSQI) (Phase II) | Start of Phase II to approximately 5 weeks
  24 item self-report measure. 19 questions are evaluated. Each item in the scale is rated between 0 (no distress) and 3 (serious distress). The total PSQI score ranges from 0-21. Sleep quality of the patients with a total score of 5 and below is considered "good". A score of greater than 5 refers to poor sleep quality.
Change in score on the Moral Injury Symptom Scale: Healthcare Professionals Version (Phase I) | Start of Phase I to approximately 2 weeks
  11 item self-report measure measuring one's experiences as a healthcare professional and how they are feeling currently. Scored between 1-10. Higher scores indicate greater moral distress.
Change in score on the Moral Injury Symptom Scale: Healthcare Professionals Version (Phase II) | Start of Phase II to approximately 5 weeks
  11 item self-report measuring one's experiences as a healthcare professional and how they are feeling currently. Scored between 1-10. Higher scores indicate greater moral distress.
Change in score on the Modified Moral Injury Events Scale (Phase I) | Start of Phase I to approximately 2 weeks
  11 item self-report measure that measures moral injury. Statements related to distress or feelings of betrayal related to potentially morally injurious events are rated on a 6 point scale ranging from 1 (strongly agree) to 6 (strongly disagree). Score range is 11-66, with higher scores reflecting greater moral injury.
Change in score on the Modified Moral Injury Events Scale (Phase II) | Start of Phase II to approximately 5 weeks
  11 item self-report measure that measures moral injury. Statements related to distress or feelings of betrayal related to potentially morally injurious events are rated on a 6 point scale ranging from 1 (strongly agree) to 6 (strongly disagree). Score range is 11-66, with higher scores reflecting greater moral injury.
Change in score on the PTSD Checklist for DSM-5 (PCL-5) (Phase I) | Start of Phase I to approximately 2 weeks
  The well-validated PCL-5 will assess self-reported PTSD symptom severity. Scores range from 0-80. Higher scores indicate greater symptom severity.
Change in score on the PTSD Checklist for DSM-5 (PCL-5) (Phase II) | Start of Phase II to approximately 5 weeks
  The well-validated PCL-5 will assess self-reported PTSD symptom severity. Scores range from 0-80. Higher scores indicate greater symptom severity.
Change in score on the Sheehan Disability Scale (SDS) (Phase I) | Start of Phase I to approximately 2 weeks
  10 point visual analog scale to rate the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms. The 3 items can be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Change in score on the Sheehan Disability Scale (SDS) (Phase II) | Start of Phase II to approximately 5 weeks
  10 point visual analog scale to rate the extent to which work/school, social life and home life or family responsibilities are impaired by his or her symptoms. The 3 items can be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Change in score on the World Health Organization Quality of Life Scale - Brief (Phase I) | Start of Phase I to approximately 2 weeks
  The minimum score is 0 and the maximum score is 100. High score shows better result.
Change in score on the World Health Organization Quality of Life Scale - Brief (Phase II) | Start of Phase II to approximately 5 weeks
  The minimum score is 0 and the maximum score is 100. High score shows better result.
Change in score on the Work and Social Adjustment Scale (WSAS) (Phase I) | Start of Phase I to approximately 2 weeks
  5 items measuring one's social functioning on items covering ability to work, home management, social leisure activities, private leisure activities, and close relationships. Each item is scored between 0-8. Lower scores are better.
Change in score on the Work and Social Adjustment Scale (WSAS) (Phase II) | Start of Phase II to approximately 5 weeks
  5 items measuring one's social functioning on items covering ability to work, home management, social leisure activities, private leisure activities, and close relationships. Each item is scored between 0-8. Lower scores are better.
Change in Score on the Occupational Stress Inventory Revised (OSI-R) (Phase I) | Start of Phase I to approximately 2 weeks
  The scale is comprised of 140 items total. The measure is comprised of 14 different scales and respondents indicate on a 5-point scale the frequency of a stress-related event.
Change in Score on the Occupational Stress Inventory Revised (OSI-R) (Phase II) | Start of Phase II to approximately 5 weeks
  The scale is comprised of 140 items total. The measure is comprised of 14 different scales and respondents indicate on a 5-point scale the frequency of a stress-related event.
Change in Score on the Multidimensional Scale of Perceived Social Support (MSPSS) (Phase I) | Start of Phase I to approximately 2 weeks
  12-item scale with a seven-point scale (from 1=strongly disagree to 7=strongly agree), resulting in a total score in the range of 12-84. Higher scores indicate higher perceived social support by Friends and Family/Significant Others.
Change in Score on the Multidimensional Scale of Perceived Social Support (MSPSS) (Phase II) | Start of Phase II to approximately 5 weeks
  12-item scale with a seven-point scale (from 1=strongly disagree to 7=strongly agree), resulting in a total score in the range of 12-84. Higher scores indicate higher perceived social support by Friends and Family/Significant Others.
Change in score on the Posttraumatic Cognitions Inventory (Phase I) | Start of Phase I to approximately 2 weeks
  33-item self-report measure is designed to assess the degree to which a participant agrees with thoughts and beliefs that have been found to be common for individuals who suffer from PTSD. The measure is rated between 1 (Totally disagree) to 7 (Totally agree). The score range is 33-231. Higher scores indicate greater symptom severity.
Change in score on the Posttraumatic Cognitions Inventory (Phase II) | Start of Phase II to approximately 5 weeks
  33-item self-report measure is designed to assess the degree to which a participant agrees with thoughts and beliefs that have been found to be common for individuals who suffer from PTSD. The measure is rated between 1 (Totally disagree) to 7 (Totally agree). The score range is 33-231. Higher scores indicate greater symptom severity.
Change in score on the Difficulties in Emotion Regulation Scale-18 (DERS-18) (Phase I) | Start of Phase I to approximately 2 weeks
  The Difficulties in Emotion Regulation Scale-18 (DERS) is a 18-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
Change in score on the Difficulties in Emotion Regulation Scale-18 (Phase II) | Start of Phase II to approximately 5 weeks
  The Difficulties in Emotion Regulation Scale-18 (DERS-18) is a 18-item self-report measure of six facets of emotion regulation. Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation.
Change in score on the Pittsburgh Insomnia Rating Scale-20 Item Version (PIRS_20) | Start of Phase I to approximately 2 weeks
  The Pittsburgh Insomnia Rating Scale is a 20 item self report measure. Items are rated on a scale from 0-3. Higher scores indicate higher insomnia severity.
Change in score on the Pittsburgh Insomnia Rating Scale-20 Item Version (PIRS_20) | Start of Phase II to approximately 5 weeks
  The Pittsburgh Insomnia Rating Scale is a 20 item self report measure. Items are rated on a scale from 0-3. Higher scores indicate higher insomnia severity.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn Difede, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CC, Difede J. A Two-Phased Telehealth Model to Treat Post-Traumatic Stress Disorder in a Health Care Worker due to the COVID-19 Pandemic: A Case Report. Telemed J E Health. 2024 Feb;30(2):601-606. doi: 10.1089/tmj.2023.0326. Epub 2023 Aug 16. PMID 37585569